CLINICAL TRIAL: NCT06589882
Title: French Prospective Cohort of Innovative Endoscopic Interventions in Expert Centers
Acronym: CoPPInE
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2024/LC-01
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Endoscopy; Innovative Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Effectiveness of diagnostic and therapeutic and/or innovative endoscopic techniques — Evaluate the effectiveness of diagnostic and therapeutic and/or innovative endoscopic techniques practiced in French expert centers over the next 10 years with the rate of technical success (procedure completed) and clinical success (cure) of the digestive pathology presented by the patient who indicated endoscopy without recourse to a new intervention (endoscopic or surgical) within 30 days of the procedure.

SUMMARY:
The creation of a multi-center French cohort pooling data from innovative endoscopies carried out in France every year would make it possible to produce excellent scientific results and analyze on a large scale the results of our current practices.

DETAILED DESCRIPTION:
Diagnostic and therapeutic digestive endoscopy has been booming over the last 10 years. Many new techniques in digestive tract or hepato-bilio-pancreatic endoscopy are introduced every year. France is the Western country with the most technical skills in terms of the number of experts relative to the size of its territory, but is lagging far behind in terms of the promotion and reimbursement of these techniques by health insurance funds. France is also experiencing difficulties in centralizing health data from the thousands of endoscopies performed in the country every year. Pooling this data across the country, following the example of certain European and international partners (the Dutch, English and Australians), would make it easier to exploit data from innovative, sometimes rare or confidential digestive endoscopy procedures, and to justify their reimbursement once their usefulness has been confirmed through large-scale descriptive prospective studies associated with national multicenter publications.

The creation of a multi-center French cohort pooling data from innovative endoscopies carried out in France every year would make it possible to produce excellent scientific results and analyze on a large scale the results of our current practi

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 yo
* Patient able to give consent
* Patient with innovative endoscopy

Exclusion Criteria:

* Opposition to participation in the present project to be notified in the file
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing innovative diagnostic or therapeutic endoscopy who do not express opposition to the use of their data from examination reports. The aim of the cohort is to provide follow-up data on innovative procedures in digestive endoscopy, in order to justify their value. Patients included in the CoPPInE innovative digestive endoscopy cohort will be considered as undergoing innovative endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2034-09-01 (Estimated); Study Completion 2034-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of diagnostic, therapeutic and/or innovative endoscopic practiced in French expert centers over the next 10 years. | 10 years

SECONDARY OUTCOMES:
Evaluate the safety of diagnostic and therapeutic and/or innovative endoscopic techniques performed in French expert centers over the next 10 years. | 10 years
Evaluate the secondary failure rate | 10 years
Evaluate operating time | 10 years
Evaluate inter-operator variability in efficacy | 10 years
Evaluate long-term efficacy | 10 years

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Nimes, Nîmes
  - Hôpital Européen Georges Pompidou AP-HP, Paris

IPD SHARING:
Plan to Share IPD: No